CLINICAL TRIAL: NCT07169084
Title: Comparison of Different Rehabilitation Approaches in Chronic Neck Pain: A Randomized Controlled Trial
Brief Title: Comparison of Different Rehabilitation Approaches in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Gamze Demircioğlu, PhD, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI-DEMIRCIOGLU-2025
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain Musculoskeletal
Keywords: Rehabilitation Approaches; Manual Therapy; Instrument-Assisted Soft Tissue Mobilization; Physical Therapy; Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy Group (Experimental): Participants receive manual therapy interventions, including posterior-anterior mobilizations, lateral glides, suboccipital release, and traction techniques based on Maitland principles.
  Interventions: Other: Manual Therapy
- Instrument-Assisted Soft Tissue Mobilization Group (Experimental): Participants receive instrument-assisted soft tissue mobilization using specialized tools on the cervical and upper thoracic regions.
  Interventions: Other: Instrument-Assisted Soft Tissue Mobilization (IASTM)

INTERVENTIONS:
Other: Manual Therapy — Manual mobilization techniques applied to the cervical and upper thoracic regions, 3 sessions/week for 4 weeks.
  Arms: Manual Therapy Group
Other: Instrument-Assisted Soft Tissue Mobilization (IASTM) — Mobilization applied with instruments to cervical and upper thoracic muscles, 3 sessions/week for 4 weeks.
  Arms: Instrument-Assisted Soft Tissue Mobilization Group

SUMMARY:
Chronic neck pain is a common musculoskeletal disorder that negatively affects daily life and quality of life. Exercise and manual therapy are widely used treatment strategies, but there is limited evidence comparing different rehabilitation approaches. This randomized controlled trial aims to compare the effects of instrument-assisted soft tissue mobilization and manual therapy on pain, functional status, cervical muscle endurance, and range of motion in individuals with chronic neck pain. Twenty-four participants will be randomly assigned to two groups and receive treatment three times per week for four weeks. Assessments will include the Visual Analog Scale, Neck Disability Index, cervical muscle endurance tests, and goniometric range of motion. The results are expected to support evidence-based strategies for managing chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years
* Diagnosis of chronic neck pain (≥12 weeks duration)
* Pain intensity ≥ 3 cm on the Visual Analog Scale (VAS)
* Voluntary participation and signed informed consent

Exclusion Criteria:

* Previous cervical spine surgery
* History of acute trauma, fracture, or dislocation in the cervical region
* Presence of neurological deficit, inflammatory disease, or systemic rheumatic condition
* Malignancy, severe cardiovascular or neurological disorder
* Participation in a similar treatment program within the past 6 months
* Current use of corticosteroids

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS), 0-10 cm (0 = no pain, 10 = worst pain imaginable) | Change from baseline to 4 weeks
  The VAS will be used to assess the intensity of neck pain. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Kâğıthane, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mylonas K, Angelopoulos P, Billis E, Tsepis E, Fousekis K. Combining targeted instrument-assisted soft tissue mobilization applications and neuromuscular exercises can correct forward head posture and improve the functionality of patients with mechanical neck pain: a randomized control study. BMC Musculoskelet Disord. 2021 Feb 21;22(1):212. doi: 10.1186/s12891-021-04080-4. PMID 33612123
- [Result] Cohen SP, Hooten WM. Advances in the diagnosis and management of neck pain. BMJ. 2017 Aug 14;358:j3221. doi: 10.1136/bmj.j3221. PMID 28807894
- [Result] Tunwattanapong P, Kongkasuwan R, Kuptniratsaikul V. The effectiveness of a neck and shoulder stretching exercise program among office workers with neck pain: a randomized controlled trial. Clin Rehabil. 2016 Jan;30(1):64-72. doi: 10.1177/0269215515575747. Epub 2015 Mar 16. PMID 25780258